CLINICAL TRIAL: NCT02968732
Title: Assessment of Reliability of Cystoscopic Evaluation Predicting pT0 Urothelial Carcinoma of the Bladder at the Time of Radical Cystectomy
Brief Title: Cystoscopic Evaluation Predicting pT0 Urothelial Carcinoma of the Bladder
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Temple University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GU-095
Record Dates: First submitted 2016-11-10; First posted 2016-11-21 (Estimated); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Surgical (Experimental)
  Interventions: Procedure: Radical Cystectomy

INTERVENTIONS:
Procedure: Radical Cystectomy

SUMMARY:
A prospective, investigational study to assess the accuracy of standardized cystoscopic evaluation with tissue sampling performed immediately prior to definitive radical cystectomy to predict pathologic tumor stage and identify patients who may benefit from bladder preservation therapy.

DETAILED DESCRIPTION:
Archival specimen of prior diagnostic TUR will be prepared as 10-20 unstained 5-10 micron slides to under-go next generation sequencing and be compared to final cystectomy specimen to investigate potential pre-treatment signatures predictive of response to chemotherapy and to understand genomic evolution of primary tumors after chemotherapy. All patients will also have urine, PBMC, and serum/plasma collected at baseline, day of procedure, 4-6 weeks post-procedure, and 6 months post-procedure. The baseline samples will be collected prior to any chemotherapy administration and prior to the procedure.

On the day of the patient's radical cystectomy, standard rigid cystourethroscopy will be performed. A urine sample will be collected from the bladder. A plasma sample will be collected while the patient is under anesthesia or in pre-op holding area. Visible tumor and prior tumor sites will be targeted for tissue sampling (no more than two sites will be targeted). A standardized tumor quantification system will be employed to document location and presence of tumor and previous biopsy sites. To this end, the investigators have developed a novel scoring system that allows for objective quantification of endoscopic findings at the time of cystoscopy and indexes presence and location of papillary tumor, erythema, and scar. Two additional random biopsies will be obtained, one from the posterior wall and one from the lateral wall for assessment of genomic signatures within normal-appearing mucosa.

Tumor location and its relationship to the ureteral orifices will be noted in order to assist the surgeon in performance of radical cystectomy. The patient will then undergo radical cystectomy as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients age >18 years at the time of consent.
2. Patients with a diagnosis of urothelial carcinoma clinical stage T1-T4NanyM0.
3. Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-3.
4. Patients must have a clinical decision to proceed with radical cystectomy by any conventional approach (open, laparoscopic, robot-assisted laparoscopic). Time from decision to surgery is usually 3-8 weeks for those who do not receive neoadjuvant chemotherapy and 10-14 weeks for those who receive neo-adjuvant chemotherapy treatment. During this time, eligibility for study participation will be verified.
5. Ability to understand and willingness to sign a written informed consent and HIPAA authorization document or a legally authorized representative who has the ability to understand and willingness to sign a written informed consent and HIPAA authorization on behalf of the participant.
6. Women of reproductive potential must have agreed to use an effective contraceptive measure.

Exclusion Criteria:

1. Patients who undergo cystectomy with non-curative intent will be excluded.
2. Patients who have undergone any prior pelvic irradiation.
3. Patients who are pregnant or nursing. Radical cystectomy and prolonged general anesthesia would place the fetus at considerable risk of demise. The prolonged recovery and debility of the patient would severely limit the patient's ability to nurse and care for an infant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the accuracy of endoscopic assessment in predicting pT0 urothelial disease in the urinary bladder at the time of radical cystectomy. | 30 days post surgery
  Endoscopic assessments will be performed using a novel scoring system that allows objective quantification of endoscopic findings at the time of cystoscopy. The findings will be compared to final pathological specimen to determine reliability of predicting pTO disease from endoscopic assessment

SECONDARY OUTCOMES:
To determine if genomic tumor signatures from pre-treatment tumor tissue can predict chemotherapy response. | up to 5years post surgery
  Archival specimen of prior diagnostic TUR will be prepared as 10-20 unstained 5-10 micron slides to under-go next generation sequencing and be compared to final cystectomy specimen to investigate potential pre-treatment signatures predictive of response to chemotherapy. Chemotherapy response will be measured by pathological assessment of residual tumor at cystectomy and graded by TNM staging criteria.
To determine how genomic tumor signatures compare before and after chemotherapy administration. | up to 5years post surgery
  Archival specimen of prior diagnostic TUR will be prepared as 10-20 unstained 5-10 micron slides to under-go next generation sequencing and be compared to final cystectomy specimen to determine genomic signatures before and after chemotherapy.
To determine if genomic signature from tissue obtained on endoscopic evaluation just prior to cystectomy can help predict final pathological stage. | up to 5years post surgery
  Comparison of baseline archival tumor tissue and final specimen will be compared for whether viable tumor tissue remains at time of surgery, for changes in total number of mutations found, whether specific mutations evolve from before to after chemo, and whether a pre-treatment genomic signature is predictive of chemo response. Specifically, DNA will be isolated from pre- and post- chemotherapy urine samples and subjected to targeted deep sequencing to support the hypothesis that mutation clearance correlates with pathologic response in the radical cystectomy specimen. These studies will provide orthogonal validation and could prove more sensitive than pathological analysis. In addition, they may serve as further basis for highly stringent selection of complete responders in whom cystectomy could be avoided in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kutikov, MD, Principal Investigator — Fox Chase Cancer Center
Locations (1):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Satyal U, Valentine H, Liu D, Slifker M, Lallas CD, Trabulsi EJ, Bukavina L, Szeto L, Hoffman-Censits JH, Mouw KW, Faltas BM, Grivas P, Ibragimova I, Porten SP, Van Allen EM, Geynisman DM, Parker DC, O'Neill JP, Drevik J, Christianson SS, Ginzburg S, Correa AF, Uzzo RG, Ross EA, Zibelman MR, Ghatalia P, Plimack ER, Kutikov A, Abbosh PH. Urine Biopsy as Dynamic Biomarker to Enhance Clinical Staging of Bladder Cancer in Radical Cystectomy Candidates. JCO Precis Oncol. 2024 Jun;8:e2300362. doi: 10.1200/PO.23.00362. PMID 38865671